CLINICAL TRIAL: NCT06968325
Title: Clinical Performance of AI-based TruRoot Designed Clear Aligner (A Randomized Clinical Trial)
Brief Title: AI-Designed Clear Aligners: A Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ahmed Abdulhussain Abbas, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1013425
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Root Resorption; Pain Perception; Treatment Duration
Keywords: Clear aligners Orthodontics Artificial intelligence Root positioning CBCT Intraoral scan TruRoot Segmentation
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-based TruRoot group (Experimental): This intervention is distinguished by its use of an AI-based treatment planning protocol that incorporates both CBCT and intraoral scan data for accurate root position estimation.
  Interventions: Device: AI-based TruRoot group:
- Conventional clear aligner group (Experimental): This intervention differs from the AI-based approach by using only intraoral scans for treatment planning, without incorporating CBCT data. Clear aligners are designed manually by experienced orthodontists based on clinical judgment and standard digital models.
  Interventions: Device: Conventional clear aligner group

INTERVENTIONS:
Device: AI-based TruRoot group: — Participants in this group will receive clear aligner treatment designed using an artificial intelligence (AI)-based system called TruRoot
  Arms: AI-based TruRoot group
Device: Conventional clear aligner group — Participants in this group will receive clear aligner treatment planned manually by expert orthodontists based only on intraoral scans.
  Arms: Conventional clear aligner group

SUMMARY:
The goal of this clinical trial is to evaluate the clinical performance and validity of applying AI-based TruRoot-designed clear aligners in adult orthodontic patients. The main questions it aims to answer are:

Do TruRoot-designed aligners achieve more accurate root positioning compared to conventional aligners?

Is there a significant difference in clinical parameters such as root resorption, pain levels, treatment duration, and occlusal outcomes between the two groups?

Is the TruRoot AI-based design a valid and clinically applicable method for planning clear aligner treatment?

Researchers will compare:

An AI-based TruRoot group, where aligners are planned using CBCT and intraoral scan superimposition to estimate true root position

A Conventional group, where aligners are designed using intraoral scans only, with expert evaluation to ensure roots remain within the alveolar bone

Participants will:

Receive clear aligner treatment based on either the TruRoot AI system or conventional planning by experts

Undergo CBCT and intraoral scans at baseline and post-treatment

Be assessed for root position accuracy, validity of AI-generated treatment plans, occlusal outcomes via the ABO Objective Grading System, root resorption, self-reported pain, and treatment duration

Attend regular follow-ups throughout the treatment period

DETAILED DESCRIPTION:
This randomized clinical trial investigates the clinical validity and performance of AI-based TruRoot-designed clear aligners compared to conventionally designed clear aligners in adult patients undergoing orthodontic treatment. The TruRoot system integrates CBCT and intraoral scan superimposition to estimate true root positioning, whereas the conventional group relies solely on intraoral scans with manual verification by expert orthodontists to ensure root positioning within the alveolar bone.

The primary aim is to assess whether AI-driven root-based treatment planning offers superior clinical outcomes in terms of root accuracy, treatment efficiency, root resorption, pain perception, and occlusal quality. Post-treatment assessments will include CBCT imaging, root position analysis, and occlusal outcome evaluation using the American Board of Orthodontics (ABO) Objective Grading System.

A comprehensive digital workflow will be applied throughout the study:

CRANEX® software will be used for generating high-resolution CBCT slice data.

BlueSky Plan or AI-based CephX® Web Viewer will be employed for segmentation and 3D modeling of dental and skeletal structures.

Clear aligner designs will be generated through BlueSky Plan software or 3Shape Clear Aligner Studio, incorporating the AI-based TruRoot protocol in the experimental group.

OnDemand 3D software will be used to evaluate root positioning within the alveolar bone post-treatment.

Geomagic® Control X™ will be utilized to quantify tooth movement and assess root volume changes throughout the treatment course.

This study will generate clinical data to validate the use of AI-powered root-based planning protocols in aligner therapy and compare them to conventional expert-driven methods

ELIGIBILITY:
Inclusion Criteria:

1. All participants should have good general health with healthy periodontium.
2. Adult patient with an age range 18-30 with fully erupted all permanent dentitions excluding third molars.
3. Skeletal and dental Cl I malocclusion with moderate crowding (little irregularity index 4-6 mm).
4. The treatment plan should be non-extraction treatment.
5. No history of trauma or root resorption

Exclusion Criteria:

1. Patients with diseases or syndromes affecting maxillofacial regions,
2. Subject with poor oral hygiene.
3. Defective and missing teeth.
4. Presence of any deep bite or open bite problems,
5. History of trauma, root resorptions and dilacerated roots.
6. Medical conditions affecting tooth movement or bone metabolism.
7. previous extraction or history of previous orthodontic treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Root position and movement | at the end of treatment
  Assessment of the accuracy of final root positions relative to the planned positions in both groups after applying certain amount of torque. and
Assessment of Root Position Relative to Alveolar Bone | before treatment begin
  Evaluation of whether the initially planned root positions in the conventional clear aligner group are contained within the alveolar bone. The assessment will be performed by importing the final STL model (planned before treatment) and superimposing it with pre-treatment CBCT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Dheaa Hussein Al-Groosh, Ph.D. Orthodontics, Study Chair — College of dentistry - University of baghdad
Locations (1):
- College of Dentistry, University of dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No